CLINICAL TRIAL: NCT03889431
Title: Community Salt Testing and Relation of Iodine Intake to Visual Information Processing of Ethiopian Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Principal Investigator, Barbara Stoecker, Regents Professor, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE1156
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Iodine Deficiency Goiter; Infant Development
MeSH Terms: interventions — Iodine; iodized salt

STUDY DESIGN:
Intervention Model Description: The mother-child dyads were randomly assigned either to receive iodine capsule (n = 53) or iodized salt (n = 53). The iodine capsule group received 225 µg of iodine daily as potassium iodide for 6 months.The iodized salt group was provided with iodized salt (30 to 40 mg iodine/kg as KIO3). One packet of salt (450 g) per household was provided starting within one week of delivery for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capsule group (Experimental): Group one received iodine capsule
  Interventions: Dietary Supplement: Iodine capsule
- Iodized salt group (Experimental): Group two received iodized salt
  Interventions: Other: Iodized Salt

INTERVENTIONS:
Dietary Supplement: Iodine capsule — 225 µg of iodine daily as a capsule of potassium iodide
  Arms: Capsule group
Other: Iodized Salt — 450 g iodized salt provided for the household weekly. Salt iodine content was 30 to 40 mg iodine /kg salt as KIO3
  Arms: Iodized salt group

SUMMARY:
This study evaluated efficacy of iodized salt for mothers and their six-month-old infants' thyroid hormones and visual information processing. Half of the participants received 450 g iodized salt for the household each week, while the other half received 225 ug iodine daily as a potassium iodide capsule.

DETAILED DESCRIPTION:
Iodine is essential for the synthesis of thyroid hormones, and thyroid hormones regulate the metabolic processes of most cells and play important roles in human growth and development. Iodine deficiency disorders can have serious consequences on brain and physical development. In neonates iodine deficiency and hence insufficient supply of thyroid hormones could cause neonatal goiter, neonatal hypothyroidism, and endemic mental retardation.

Iodine deficiency disorders can be prevented and controlled by providing iodine and iodine can be provided in different ways. However, the United Nations Children's Fund and the World Health Organization jointly recommended salt iodization where iodized salt is accessible. Iodized salt is a safe, cost effective and sustainable strategy to ensure sufficient intake of iodine by all individuals and to improve maternal and infant health. However, although the effect of iodine on human health is well established efficacy of iodized salt has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* The women must be lactating and must have an infant less than or equal to one week old.
* Mothers had to volunteer to participate in the study.

Exclusion Criteria:

* Any hyperthyroidism symptoms manifested by nervousness, anxiety, heart palpitations, or rapid pulse.
* If infants had fever, cough or severe (>3/day) diarrhea
* Any allergic reaction such as acne, weakness, or foul breath

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2013-01-30 (Actual); Study Completion 2013-08-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline breast milk iodine concentration (µg/L) at six months | First week after delivery and at six months
  Laboratory analysis
Change from baseline urinary iodine concentration (µg/L at six months | First week after delivery and at six months
  Laboratory analysis
Change from baseline Infants' anthropometric measurement (Z-score) at six months | First week after delivery and at six months
  Measurement

SECONDARY OUTCOMES:
Change from baseline thyroid hormones status at six months | First week after delivery and at six months
  Laboratory analysis
Infants' visual information processing | At six months after delivery
  Looking behavior test

CONTACTS AND LOCATIONS:
Overall Officials: Tafere Gebreegziabher, PhD, Principal Investigator — Central Washington University & Hawassa University
Locations (1):
- Hawassa University, Awasa, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan S, Kilby MD. Thyroid hormone and central nervous system development. J Endocrinol. 2000 Apr;165(1):1-8. doi: 10.1677/joe.0.1650001. No abstract available. PMID 10750030
- [Result] Zimmermann MB. The effects of iodine deficiency in pregnancy and infancy. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1:108-17. doi: 10.1111/j.1365-3016.2012.01275.x. PMID 22742605
- [Result] Zimmermann MB. The Importance of Adequate Iodine during Pregnancy and Infancy. World Rev Nutr Diet. 2016;115:118-24. doi: 10.1159/000442078. Epub 2016 May 19. PMID 27198746
- [Result] Dold S, Zimmermann MB, Jukic T, Kusic Z, Jia Q, Sang Z, Quirino A, San Luis TOL, Fingerhut R, Kupka R, Timmer A, Garrett GS, Andersson M. Universal Salt Iodization Provides Sufficient Dietary Iodine to Achieve Adequate Iodine Nutrition during the First 1000 Days: A Cross-Sectional Multicenter Study. J Nutr. 2018 Apr 1;148(4):587-598. doi: 10.1093/jn/nxy015. PMID 29659964
- [Result] Robinson SM, Crozier SR, Miles EA, Gale CR, Calder PC, Cooper C, Inskip HM, Godfrey KM. Preconception Maternal Iodine Status Is Positively Associated with IQ but Not with Measures of Executive Function in Childhood. J Nutr. 2018 Jun 1;148(6):959-966. doi: 10.1093/jn/nxy054. PMID 29767745
- [Result] Vongchana M, Ounjaijean S, Tongsong T, Traisrisilp K. The effectiveness of iodine supplementation during pregnancies in geographical areas of high prevalence of iodine insufficiency. J Obstet Gynaecol. 2018 Aug;38(6):756-761. doi: 10.1080/01443615.2017.1410534. Epub 2018 Mar 12. PMID 29526129
- [Result] WHO Secretariat; Andersson M, de Benoist B, Delange F, Zupan J. Prevention and control of iodine deficiency in pregnant and lactating women and in children less than 2-years-old: conclusions and recommendations of the Technical Consultation. Public Health Nutr. 2007 Dec;10(12A):1606-11. doi: 10.1017/S1368980007361004. No abstract available. PMID 18053287
- [Result] Zimmermann MB. Iodine deficiency in pregnancy and the effects of maternal iodine supplementation on the offspring: a review. Am J Clin Nutr. 2009 Feb;89(2):668S-72S. doi: 10.3945/ajcn.2008.26811C. Epub 2008 Dec 16. PMID 19088150
- [Result] Vejbjerg P, Knudsen N, Perrild H, Carle A, Laurberg P, Pedersen IB, Rasmussen LB, Ovesen L, Jorgensen T. Effect of a mandatory iodization program on thyroid gland volume based on individuals' age, gender, and preceding severity of dietary iodine deficiency: a prospective, population-based study. J Clin Endocrinol Metab. 2007 Apr;92(4):1397-401. doi: 10.1210/jc.2006-2580. Epub 2007 Jan 30. PMID 17264188
- [Result] Gebreegziabher T, Stoecker BJ. Comparison of two sources of iodine delivery on breast milk iodine and maternal and infant urinary iodine concentrations in southern Ethiopia: A randomized trial. Food Sci Nutr. 2017 Apr 7;5(4):921-928. doi: 10.1002/fsn3.477. eCollection 2017 Jul. PMID 28748081
- [Result] Kennedy T, Thomas DG, Woltamo T, Abebe Y, Hubbs-Tait L, Sykova V, Stoecker BJ, Hambidge KM. Growth and Visual Information Processing in Infants in Southern Ethiopia. J Appl Dev Psychol. 2008 Mar 1;29(2):129-140. doi: 10.1016/j.appdev.2007.12.003. PMID 19684873
- [Result] Reynolds GD. Infant visual attention and object recognition. Behav Brain Res. 2015 May 15;285:34-43. doi: 10.1016/j.bbr.2015.01.015. Epub 2015 Jan 14. PMID 25596333
- [Result] Santiago P, Velasco I, Muela JA, Sanchez B, Martinez J, Rodriguez A, Berrio M, Gutierrez-Repiso C, Carreira M, Moreno A, Garcia-Fuentes E, Soriguer F. Infant neurocognitive development is independent of the use of iodised salt or iodine supplements given during pregnancy. Br J Nutr. 2013 Sep 14;110(5):831-9. doi: 10.1017/S0007114512005880. Epub 2013 Feb 4. PMID 23375074
- [Result] Velasco I, Carreira M, Santiago P, Muela JA, Garcia-Fuentes E, Sanchez-Munoz B, Garriga MJ, Gonzalez-Fernandez MC, Rodriguez A, Caballero FF, Machado A, Gonzalez-Romero S, Anarte MT, Soriguer F. Effect of iodine prophylaxis during pregnancy on neurocognitive development of children during the first two years of life. J Clin Endocrinol Metab. 2009 Sep;94(9):3234-41. doi: 10.1210/jc.2008-2652. Epub 2009 Jun 30. PMID 19567536
- [Result] Delange F. Iodine requirements during pregnancy, lactation and the neonatal period and indicators of optimal iodine nutrition. Public Health Nutr. 2007 Dec;10(12A):1571-80; discussion 1581-3. doi: 10.1017/S1368980007360941. PMID 18053281
- [Result] Bouhouch RR, Bouhouch S, Cherkaoui M, Aboussad A, Stinca S, Haldimann M, Andersson M, Zimmermann MB. Direct iodine supplementation of infants versus supplementation of their breastfeeding mothers: a double-blind, randomised, placebo-controlled trial. Lancet Diabetes Endocrinol. 2014 Mar;2(3):197-209. doi: 10.1016/S2213-8587(13)70155-4. Epub 2013 Nov 22. PMID 24622750
- [Result] Antonangeli L, Maccherini D, Cavaliere R, Di Giulio C, Reinhardt B, Pinchera A, Aghini-Lombardi F. Comparison of two different doses of iodide in the prevention of gestational goiter in marginal iodine deficiency: a longitudinal study. Eur J Endocrinol. 2002 Jul;147(1):29-34. doi: 10.1530/eje.0.1470029. PMID 12088916
- [Result] Rohner F, Zimmermann M, Jooste P, Pandav C, Caldwell K, Raghavan R, Raiten DJ. Biomarkers of nutrition for development--iodine review. J Nutr. 2014 Aug;144(8):1322S-1342S. doi: 10.3945/jn.113.181974. Epub 2014 Jun 25. PMID 24966410
- [Result] Ghirri P, Lunardi S, Boldrini A. Iodine supplementation in the newborn. Nutrients. 2014 Jan 20;6(1):382-90. doi: 10.3390/nu6010382. PMID 24448111
- [Result] Taylor RM, Fealy SM, Bisquera A, Smith R, Collins CE, Evans TJ, Hure AJ. Effects of Nutritional Interventions during Pregnancy on Infant and Child Cognitive Outcomes: A Systematic Review and Meta-Analysis. Nutrients. 2017 Nov 20;9(11):1265. doi: 10.3390/nu9111265. PMID 29156647